CLINICAL TRIAL: NCT02743845
Title: Gene Discovery Core, The Manton Center
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alan H. Beggs, Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 10-02-0053
Record Dates: First submitted 2016-01-04; First posted 2016-04-19 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Undiagnosed Conditions; Rare Disorders; Orphan Diseases
Keywords: Rare; Undiagnosed; Orphan Disease; Genomic Sequencing
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA RNA Tissue Samples Cell lines
Oversight: Data Monitoring Committee: No

SUMMARY:
The Gene Discovery Core at The Manton Center for Orphan Disease Research based at Boston Children's Hospital studies families with rare, poorly understood or undiagnosed, but suspected genetic conditions. The primary goal of the research is to better understand the genes and proteins (gene products) involved in rare diseases. The researchers hope that our studies will allow for improved diagnosis and treatment of individuals with rare disease in the future. Individuals with any rare/undiagnosed condition are eligible to enroll.

Enrollment includes:

* Providing DNA and tissue samples (when available)
* Access to participants' medical records
* Access to genomic data (when available)

Samples are used for genetic analysis (primarily exome and genome sequencing or reanalysis) to identify the genetic cause for the individual's illness. Individual research results are returned to families through their health care provider after confirmation in a clinical lab. If a cause is identified, that can be reported back to the family through their health care provider and the study's genetic counselor. When possible, the investigators also collect samples from parents and full-siblings as well as any other affected family members.

DETAILED DESCRIPTION:
Participants may be recruited from Boston Children's Hospital (BCH) or from off-site collaborators/healthcare providers who determine a participant as eligible. Participants may also contact the lab directly after hearing about the research through other individuals, recruitment materials, or the study's website (www.childrenshospital.org/mantoncenter). After consenting to participation, individuals with rare disorders with a suspected, but unknown/poorly understood genetic basis, and their family members are asked to participate in the study by providing 1) relevant medical information/records and family history 2) a blood/saliva/DNA/RNA sample, and 3) preexisting tissue samples (including preexisting prenatal samples) that is no longer needed for clinical care (if available) or future tissue sample specifically for research purposes.

The medical records and family history allow the investigators to gain a better understanding of the specific disease symptoms seen in an individual or family. The blood/saliva sample is used to obtain DNA and/or RNA, and/or other biochemical which can then be analyzed for identifying the genetic bases of disease pathophysiology using various approaches including genomic sequencing. Tissue samples obtained from individual participants are employed to better understand gene expression and protein interactions through investigations such as (but not limited to) immunohistochemical and microarray analysis.

This study project will be ongoing for an indefinite period of time, and participation is continuous unless an individual requests to be removed from the study. Participants can request to withdraw at any time. Active participation primarily takes place at the time of enrollment and on a case-by-case basis thereafter for providing clinical updates and/or additional samples. Risks include those associated with routine blood draws/saliva sample collections and emotional distress associated with genetic and/or medical research. Risks are minimized as much as possible by an open consent process and privacy/confidentiality safeguards, including a certificate of confidentiality from the NIH and the use of de-identified, numerical codes to refer to participants with collaborators. Although there are no immediate, direct benefits to participants, the possible benefits of this study include the development of new diagnostic tests and more detailed prognostic information for participants and their families. In addition, this study may lead to a better understanding of the pathophysiology of these conditions, leading to the development of treatments and cures for both rare and more common disorders in the future.

ELIGIBILITY:
Inclusion Criteria:

* Having a known or uncertain rare diagnosis which may have a poorly understood genetic component and/or be a relative to a person with such a diagnosis

Exclusion Criteria:

* Not having such a diagnosis and/or not being related to such an individual

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a rare or unknown but presumed genetic diagnosis and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-02; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of rare or novel disease-causing genetic variants for a participant's disorder | 1-10 years
  Functional analysis, including animal modeling and cell line assays, will be performed for novel candidate genes. When a molecular diagnosis is identified for a family, this is reported back through a designated health care provider.
Characterization of clinical features of novel and rare disorders using Human Phenotype Ontology (HPO) terms | 1-10 years
  As known and new disease genes are identified the resulting genotypes are correlated with subject phenotypes.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
If a genetic etiology is found, individual results are reported back to families.